CLINICAL TRIAL: NCT03919357
Title: Assessment of the Diagnostic Approach to Specific Language Disorders and Learning Using a New Calibrated Tool: the Modular Battery Tests Computerized (BMTi)
Brief Title: Using a New Calibrated Tool in Specific Language and Learning Disorders : the BMTi
Acronym: ValidBMTI
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Collaborators: Association pour la recherche des troubles de l'apprentissage (Unknown); Orthoédition (Unknown); Association Française de Pédiatrie Ambulatoire- AFPA (Unknown); Association pour l'Etude du Développement de l'Enfant (Unknown)
Responsible Party: Sponsor
Other Study IDs: ValidBMTI2018; 2018-A01870-55 (Other: ID-RCB)
Record Dates: First submitted 2019-04-04; First posted 2019-04-18 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Learning Disorders, Specific; Developmental Disability
MeSH Terms: conditions — Specific Learning Disorder; Developmental Disabilities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Verbal: Passing of a specialized questionnaire on verbal disorders
  Interventions: Behavioral: BMT-i
- Non-verbal: Passing of a specialized questionnaire on non verbal disorders
  Interventions: Behavioral: BMT-i
- Attention: Passing of a specialized questionnaire on attention disorders
  Interventions: Behavioral: BMT-i
- Complaint about learning: Passing of a specialized questionnaire on learning disorders
  Interventions: Behavioral: BMT-i

INTERVENTIONS:
Behavioral: BMT-i — Passing the BMT-i test

SUMMARY:
The group of experts at HAS has defined the places of first and second-line workers in specific disorders of development and learning, as defined in the international diagnostic classifications International Classification of Diseases (CIM) CIM 11 and Diagnostic and Statistical Manual of Mental Disorders (DSM) DSM 5. The referral to a second-level structure, a multidisciplinary structure in charge of carrying out the different cognitive assessments, requires a preliminary evaluation.

This orientation is based on a medical consultation, carried out by a doctor specialized in the field, with an exploration tool adapted to the different fields concerned.

The BMTi, a battery of third-generation tests (after the Rapid battery of evaluation of the cognitive functions (BREV) and then the Evaluation of cognitive functions and learning of the child (EDA)) will enable the doctor, from 2018, to carry out this orientation in a relevant way in response to children with a complaint about neurodevelopment and learning. .

The research project aims to validate this hypothesis, by comparing the diagnoses posed in a conventional way with the various multidisciplinary assessments, with the results of the transfer of all or part of the subtests of the BMTi by a doctor of second resort.

DETAILED DESCRIPTION:
The group of experts at High Authority of Health (HAS) has defined the places of first and second-line workers in specific disorders of development and learning, as defined in the international diagnostic classifications CIM 11 and DSM 5. The referral to a second-level structure, a multidisciplinary structure in charge of carrying out the different cognitive assessments, requires a preliminary evaluation.

This orientation is based on a medical consultation, carried out by a doctor specialized in the field, with an exploration tool adapted to the different fields concerned.

The BMTi, a battery of third-generation tests (after the BREV and then the EDA) will enable the doctor, from 2018, to carry out this orientation in a relevant way in response to children with a complaint about neurodevelopment and learning. .

The research project aims to validate this hypothesis, by comparing the diagnoses posed in a conventional way with the various multidisciplinary assessments, with the results of the transfer of all or part of the subtests of the BMTi by a doctor of second resort.

This research project finds its place in a more global approach for a complete application of the recommendations of the group of experts of the High Authority of Health with:

* the systematic evaluation of educational prevention strategies by intensive training in small groups of children with similar needs, in schools,
* the evaluation of the role of the primary care physician in the prescription of the initial investigation report in the face of a simple reading, writing or numeracy disorder (research project with letter of intent filed in the framework of the call for tenders 38/5000 general direction of the offer of care (DGOS) PREPS 2018),
* the current project to validate referral tools to second-level appraisals,
* an evaluation project of the financing modalities filed under the regional health agency "Occitanie" in the framework of the call for tenders of article 51,
* the introduction of training courses for the first and second-line tools for ambulatory doctors.

ELIGIBILITY:
Inclusion Criteria:

* Child aged 5 to 13
* Complex complaint affecting one of the different areas of development and learning
* Affiliation to a social security scheme

Exclusion Criteria:

* Diagnosis of intellectual development disorder of autism spectrum disorder and suspect or confirm
* Refusal to participate

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children between 5 and 13 years old with a complex developmental and learning disorder
Sampling Method: Non-Probability Sample
Enrollment: 229 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity of BMT-i (modular computerized test battery) | 3 months
  Calculation of the sensitivity of the BMT-i compared to the reference balance sheets
Specificity of BMT-i | 3 months
  Calculation of the specificity of the BMT-i compared to the reference balance sheets

SECONDARY OUTCOMES:
Sensitivity and specificity of the BMT-i by type of complaint | 3 months
  Calculation of the sensitivity and specificity of the BMT-i compared to the reference balance in each type of complaint (oral language, learning, graphics and attention)
Kappa de Cohen test between BMTi assessments and the reference assessments | 3 months
  Assessment of the concordance between the BMTi assessments and the baseline assessments
Concordance between investigators evaluations and reviewers evaluations | 3 months
  Evaluation of the concordance between the BMTi evaluations rated by the investigators and the reviewers
Curves ROC (Receiver operating characteristic) | 3 months
  Receiver operating characteristic (ROC) curves to validate selected BMT-i diagnostic thresholds

CONTACTS AND LOCATIONS:
Locations (16):
- France (15):
  - Cabinet du Dr Vurpillat-Almanza, Besançon
  - Cabinet du Dr Piollet, Chamalières
  - Cabinet du Dr Gelbert, Chambéry
  - CH Versailles - André Mignot, Le Chesnay
  - Centre Médical Pédiatrique Flammarion, Marseille
  - Hôpital Saint Eloi - Montpellier, Montpellier
  - Cabinet du Dr Kochert, Orléans
  - Centre Paris Santé Réussite, Paris
  - Cabinet du Dr Cahn-Sellem, Puteaux
  - CHU de Rouen, Rouen
  - Cabinet du Dr Reynaud, Saint-Denis
  - Cabinet du Dr Willig, Toulouse
  - Cabinet du Dr Pineau, Trélazé
  - Cabinet du Dr Lubelski, Verrières-le-Buisson
  - Cabinet du Dr Werner, Villeneuve-lès-Avignon
- Cabinet du Dr Dulorme, Le Lamentin, Martinique

IPD SHARING:
Plan to Share IPD: No